CLINICAL TRIAL: NCT02142309
Title: Effect of Glimepiride, Vildagliptin, Pioglitazone and Canagliflozin on Durability of Glycemic Control After Metformin Failure in Type 2 Diabetes
Brief Title: Glycemic Durability After Metformin Failure
Acronym: AMAZING
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Dario Giugliano, Full Prof of Endocrinology and Metbaolism, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGM 7-2006
Record Dates: First submitted 2014-04-26; First posted 2014-05-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Vildagliptin; Pioglitazone; Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glimepiride (Experimental): up to 4 mg/day
  Interventions: Drug: Glimepiride
- Vildagliptin (Experimental): 50 mg bid
  Interventions: Drug: Vildagliptin
- Pioglitazone (Experimental): up to 30 mg/day
  Interventions: Drug: Pioglitazone
- Canagliflozin (Experimental): 300 mg/day
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Glimepiride — Weekly adjustment based on self-monitoring of blood glucose level to a maximum of 4 mg daily
  Arms: Glimepiride
Drug: Vildagliptin — Reduce to 50 mg if estimated glomerular filtration rate (eGFR) <45 mL/min
  Arms: Vildagliptin
Drug: Pioglitazone — Start with 15 mg/day and advance to 30 mg/day
  Arms: Pioglitazone
Drug: Canagliflozin — Start with 200 mg/day and advance to 300 mg/day on the basis of fasting glucose monitoring
  Arms: Canagliflozin

SUMMARY:
Type 2 diabetes is epidemic and its treatment has become more and more difficult. Consensus algorithms have been developed to help clinicians to select among the numerous medications and their combinations for achieving and maintaining a target glycated hemoglobin A1c (HbA1c) of <7%.

AMAZING, a pragmatic clinical trial, aims to compare commonly used oral diabetes medications, when combined with metformin, on glycemia-lowering effectiveness.

DETAILED DESCRIPTION:
* Source data verification: paper or electronic medical records.
* Statistical analysis: All analyses will compare the randomly assigned treatment groups under the intention- to-treat principle

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed, type 2 diabetic patients, failing to diet

Exclusion Criteria:

* Suspected type 1 diabetes or secondary diabetes resulting from specific causes
* Current or previous (within past 3 months) treatment with any investigational drug
* Any major cardiovascular event in previous year
* Plans for pregnancy during the course of the study for women of childbearing potential
* Serum creatinine level >1.3 mg/dL in women and >1.4 mg/dL in men
* History of cancer, other than nonmelanoma skin cancer, that required therapy in the 5 years before randomization
* Treatment with oral, loal, systemic glucocorticoids 14. Treatment with atypical antipsychotics

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2005-10; Primary Completion 2015-10 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is maintenance of metabolic control (glycemic durability), defined as time to primary failure with a HbA1c value >7% on maximally tolerated doses of the assigned drug. | Six years

SECONDARY OUTCOMES:
Continuous glucose monitoring for 72 consecutive hours at least once each year of follow-up | 6 years

OTHER OUTCOMES:
Changes of low density lipoprotein cholesterol level from baseline each year of follow up | 6 years
Changes of high density lipoprotein cholesterol level from baseline each year of follow up | six years
Changes of triglyceride level from baseline each year of follow up | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD PHD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (2):
- Italy (2):
  - Katherine Esposito, Naples, Naples
  - Department of Geriatrics and Metabolic Diseases, Naples